CLINICAL TRIAL: NCT00155480
Title: Establish Finite Element Mesh of the Numerical Models of the Thoracic Aorta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461700626
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Heart Diseases
Keywords: thoracic aorta; finite element mesh
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Procedure: computed tomography

SUMMARY:
This study will be using finite element meshes and averaged algorithms to create the numerical thoracic aorta at different ages.

DETAILED DESCRIPTION:
This study will be using finite element meshes and averaged algorithms to create the numerical thoracic aorta at different ages.

ELIGIBILITY:
Inclusion Criteria:

* Normal thoracic aorta

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2000-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy

SECONDARY OUTCOMES:
sensitivity
specificity

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Jye Chen, MD, PhD, Principal Investigator — Dept. Medical Imaging, NTaiwanUH
Locations (1):
- Dept. of Medical Imaging, NTaiwanUH, Taipei, Taiwan